CLINICAL TRIAL: NCT01242839
Title: Randomized Multicentric Double Blinded Study Evaluating CACICOL20 Efficiency Versus Placebo Corneal Chronic Ulcers Healing
Brief Title: Randomized Double Blinded Study Evaluating CACICOL20 Efficiency Versus Placebo Corneal Chronic Ulcers Healing
Acronym: UNICOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organ, Tissue, Regeneration, Repair and Replacement (Industry)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT08L06UC
Record Dates: First submitted 2010-09-03; First posted 2010-11-17 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Corneal Ulcer
Keywords: CACICOL20
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CACICOL20 (Experimental): Arm that receives CACICOL20 treatment each 2 days for 3 months/until closure of the ulcer
  Interventions: Device: CACICOL20
- Placebo (Placebo Comparator): The placebo is applicated each 2 days on patient cornea for 3 months/ until ulcer closure.
  Interventions: Device: Placebo
- CACICOL20 and Placebo (Experimental): Patient applies the treatment each 2 days for 3 months or until closure of the ulcer. This treatment is alternatively CACICOL20 or Placebo : so the patient receives CACICOL20 each 4 days. CACICOL20 and placebo strips are strictly similar and cannot be identified.
  Interventions: Device: CACICOL20

INTERVENTIONS:
Device: CACICOL20 — CACICOL20 is a solution of dextran & poly(carboxymethylglucose sulphate)in physiological salt serum. CACICOL20 is presented in 0.33 mL strip. One drop is instilled at each application to impregnate cornea.
  Arms: CACICOL20; CACICOL20 and Placebo
Device: Placebo — It is the placebo of CACICOL20, containing dextran in physiological serum salt. It is presented, like CACICOL20, in a 0.33 mL strip. One drop is delivered at each application.
  Arms: Placebo

SUMMARY:
CACICOL20 is a biodegradable nanopolymer engineered to mimic glycosaminoglycans such as heparan sulfates. Applied to the corneal lesion, it replaces damaged heparan sulfates in the matrix scaffold. CACICOL20 binds to matrix proteins such as collagen and cytokines or endogenous growth factors of the cellular microenvironment. CACICOL20 provides a protective function and restores the matrix architecture. This produces a suitable spatial environment for cells to respond properly to the cascade of signals needed for tissue regeneration to resume.

The ophthalmic solution, CACICOL20, used for corneal ulcers is very well tolerated both locally and generally, as proved by a pilot study which as been conducted at the "Hôpital des XV-XX" in Paris (France). It reduces the pain significantly and increases corneal ulcer healing (all ulcers treated were resistant to all other usual therapies).

Therefore, the accuracy of a Randomized multicentric double blinded study to evaluate the efficacy of CACICOL20 versus placebo for chronic corneal ulcer healing has been shown and will begin mid-may 2010. In this study, CACICOL20 will be applied every 2 or 4 days for 3 months.

The aim of the study is a double blinded comparison of complete chronic corneal ulcers healing rate within 3 months in 3 groups of patient double blinded randomized between CACICOL20 instillations distribution and physiological salt solution instillations distribution.

The main judgment criteria is healing rate within 3 months defined as corneal ulcer complete closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-infectious, corneal chronic ulcer, painful or not ,whose depth does not exceed the superficial stroma.
* Resistance of corneal pathology to standard treatment: eye drops to promote healing, tear substitutes, anti-inflammatory drugs, cyclosporin.
* Patients previously treated for the corneal pathology, assessed ineffective or Insufficiently effective by the investigator
* Patients using wetting gel or eye drops without conservator during the inclusion
* Anti-inflammatory local treatments must be stopped for at least 8 days.
* No contact lenses or lenses must be removed for at least 8 days.
* Age of inclusion ≥ 18 years.
* Written and signed informed consent from patient.
* Realization of a preliminary medical examination.
* Covers by social insurance

Exclusion Criteria:

* Ulcers deeper than the superficial stroma, perforated ulcers or pre-perforated
* Corneal abscess
* Infectious and progressive ulcerative keratitis
* Patients receiving anti-inflammatory eye drops or steroid with cyclosporine treatment (in this case, possibility of inclusion in the clinical protocol after a Case "wash-out of 8 days)
* Patients on long-term eye drops containing preservatives and can not be stopped or replaced by an equivalent without preservatives
* Patients on systemic anti-inflammatory, anti-allergic, psychotropic or antibiotics therapies, modified since less than 10 days or likely to be on short-term
* Wearing contact lenses if patient has not been stopped at least eight days before the start of the protocol
* ocular surgery within the last 3 months
* patient already included in another clinical trial with an investigational product
* Pregnant patients or breastfeeding
* Person under a legal protection measure, under guardianship
* Unable to follow up medical examinations for geographical, social or psychological reasons
* Not cover by social insurance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Healing rate | Within 1 months
  The main judgment criteria is healing rate within 3 months defined as corneal ulcer complete closure.

SECONDARY OUTCOMES:
Healing rate | 2 and 3 months
  Complete Healing rate of the ulcer at 1 and 2 months defined as corneal ulcer complete closure, the evaluation of the pain with visual pain scale and evaluation of the quotation of analgesic treatments used by the patient.
Visual pain scale | 1, 2 and 3 months
  Complete Healing rate of the ulcer at 1 and 2 months defined as corneal ulcer complete closure, the evaluation of the pain with visual pain scale and evaluation of the quotation of analgesic treatments used by the patient.
Associated treatments quotation | 1, 2 and 3 months
  Quotation of analgesic treatments used and assessment of the effects of lubricant eye drops on the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Baudouin, MD, Principal Investigator — XV- XX Hospital - Paris
Locations (21):
- France (21):
  - Centre Hospitalier Universitaire Amiens, Amiens
  - CHU Angers, Angers
  - Hopital Avicennes, Bobigny
  - Centre Hospitalier Ambroise Paré, Boulogne-Billancourt
  - Hôpital Gabriel Montpied - CHU Clermont Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Hôpital BICETRE, Le Kremlin-Bicêtre
  - CHRU Lille Hôpital Huriez, Lille
  - CHU Limoges, Hôpital Dupuytren, Limoges
  - CHU LYON, Hôpital Edouard Herriot, Lyon
  - AP-HM Hôpital de la Timone, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - AP-HP Hôpital Hôtel-Dieu, Paris
  - Centre Hospitalier des Quinze Vingt, Paris
  - Hôpital BICHAT - CLAUDE-BERNARD, Paris
  - CHU Hopitaux de Rouen, Rouen
  - Centre Hospitalier Universitaire de Saint-Etiennne, Saint-Etienne
  - CH Saint Louis, Saint Jean d'Angély, Saint-Jean-d'Angély
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire de Tours, Tours